CLINICAL TRIAL: NCT01132495
Title: Fractional Flow Reserve-Guided Percutaneous Coronary Intervention Plus Optimal Medical Treatment Versus Optimal Medical Treatment Alone in Patients With Stable Coronary Artery Disease
Brief Title: FAME II - Fractional Flow Reserve (FFR) Guided Percutaneous Coronary Intervention (PCI) Plus Optimal Medical Treatment (OMT) Verses OMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0904
Record Dates: First submitted 2010-05-20; First posted 2010-05-28 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: Stable angina; angina pectoris; PCI; FAME; FAME II; FFR; Fractional Flow Reserve; Pressure wire
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina Pectoris | interventions — Stents; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A: PCI plus OMT (Other): PCI plus optimal medical treatment
  Interventions: Other: Stenting plus OMT
- Cohort A: OMT alone (Other): Optimal medical treatment alone
  Interventions: Other: OMT
- Cohort B (Other): FFR > 0.80; treatment according to local practice
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Stenting plus OMT — FFR guided PCI, plus OMT
  Arms: Cohort A: PCI plus OMT
Other: OMT — OMT alone
  Arms: Cohort A: OMT alone
Other: Standard of care — FFR > 0.80; treatment according to local practice
  Arms: Cohort B

SUMMARY:
The overall purpose of the FAME II trial is to compare the clinical outcomes, safety and cost-effectiveness of FFR-guided PCI plus optimal medical treatment (OMT) versus OMT alone in patients with stable coronary artery disease.

DETAILED DESCRIPTION:
Prospective, multi-center, multi-national, multi-continental, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with

   * stable angina or,
   * stabilized angina pectoris or,
   * atypical chest pain or no chest pain but with documented silent ischemia
2. at least one stenosis is present of at least 50% in one major native epicardial coronary artery and supplying viable myocardium
3. Eligible for PCI
4. Signed written informed consent

Exclusion Criteria:

1. Patients in whom the preferred treatment is CABG
2. Patients with left main coronary artery disease requiring revascularization
3. Patients with a recent STEMI or Non-STEMI
4. Prior CABG
5. Contra-indication to dual antiplatelet therapy
6. LVEF < 30%
7. Severe LV hypertrophy
8. Planned need for concomitant cardiac surgery
9. Extremely tortuous or calcified coronary arteries precluding FFR measurements
10. A life expectancy of less than 2 years
11. Age under 21

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard De Bruyne, MD, Principal Investigator — O.L.Vrouwzlekenhuis Hospital
Locations (29):
- United States (6):
  - VA Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Tulane University, New Orleans, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
- OLV Ziekenhuis, Aalst, Belgium
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- Czechia (2):
  - Masaryk University and University Hospital Brno, Brno
  - Na Homolce Hospital, Prague
- Rigshospitalet University Hospital, Copenhagen, Denmark
- Hospices Civils de Lyon, Bron, France
- Germany (3):
  - Heart Center Leipzig, Leipzig
  - Klinikum der Universitat Munchen, München
  - Stadtisches Klinikum Munchen, München
- Gottsegen Hungarian Institute of Cardiology, Budapest, Hungary
- Azienda Ospedaliero Universitaria de Ferrara, Ferrara, Italy
- Netherlands (3):
  - Catharina-Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
  - Isala Klinieken, Zwolle
- Clinical Center Kragujevac, Kragujevac, Serbia
- Sweden (2):
  - Orebro University Hospital, Örebro
  - Sodersjukhuset AB, Stockholm
- United Kingdom (5):
  - Royal Victoria Hospital, Belfast
  - Edinburgh Heart Centre, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Kings College Hospital, London
  - Southampton University Hospitals NHS, Southampton

REFERENCES:
- [Derived] Nishi T, Piroth Z, De Bruyne B, Jagic N, Mobius-Winkler S, Kobayashi Y, Derimay F, Fournier S, Barbato E, Tonino P, Juni P, Pijls NHJ, Fearon WF. Fractional Flow Reserve and Quality-of-Life Improvement After Percutaneous Coronary Intervention in Patients With Stable Coronary Artery Disease. Circulation. 2018 Oct 23;138(17):1797-1804. doi: 10.1161/CIRCULATIONAHA.118.035263. PMID 30354650
- [Derived] Xaplanteris P, Fournier S, Pijls NHJ, Fearon WF, Barbato E, Tonino PAL, Engstrom T, Kaab S, Dambrink JH, Rioufol G, Toth GG, Piroth Z, Witt N, Frobert O, Kala P, Linke A, Jagic N, Mates M, Mavromatis K, Samady H, Irimpen A, Oldroyd K, Campo G, Rothenbuhler M, Juni P, De Bruyne B; FAME 2 Investigators. Five-Year Outcomes with PCI Guided by Fractional Flow Reserve. N Engl J Med. 2018 Jul 19;379(3):250-259. doi: 10.1056/NEJMoa1803538. Epub 2018 May 22. PMID 29785878
- [Derived] Ciccarelli G, Barbato E, Toth GG, Gahl B, Xaplanteris P, Fournier S, Milkas A, Bartunek J, Vanderheyden M, Pijls N, Tonino P, Fearon WF, Juni P, De Bruyne B. Angiography Versus Hemodynamics to Predict the Natural History of Coronary Stenoses: Fractional Flow Reserve Versus Angiography in Multivessel Evaluation 2 Substudy. Circulation. 2018 Apr 3;137(14):1475-1485. doi: 10.1161/CIRCULATIONAHA.117.028782. Epub 2017 Nov 21. PMID 29162610
- [Derived] Fearon WF, Nishi T, De Bruyne B, Boothroyd DB, Barbato E, Tonino P, Juni P, Pijls NHJ, Hlatky MA; FAME 2 Trial Investigators. Clinical Outcomes and Cost-Effectiveness of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention in Patients With Stable Coronary Artery Disease: Three-Year Follow-Up of the FAME 2 Trial (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation). Circulation. 2018 Jan 30;137(5):480-487. doi: 10.1161/CIRCULATIONAHA.117.031907. Epub 2017 Nov 2. PMID 29097450
- [Derived] Barbato E, Toth GG, Johnson NP, Pijls NH, Fearon WF, Tonino PA, Curzen N, Piroth Z, Rioufol G, Juni P, De Bruyne B. A Prospective Natural History Study of Coronary Atherosclerosis Using Fractional Flow Reserve. J Am Coll Cardiol. 2016 Nov 29;68(21):2247-2255. doi: 10.1016/j.jacc.2016.08.055. PMID 27884241
- [Derived] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Derived] Fearon WF, Shilane D, Pijls NH, Boothroyd DB, Tonino PA, Barbato E, Juni P, De Bruyne B, Hlatky MA; Fractional Flow Reserve Versus Angiography for Multivessel Evaluation 2 (FAME 2) Investigators. Cost-effectiveness of percutaneous coronary intervention in patients with stable coronary artery disease and abnormal fractional flow reserve. Circulation. 2013 Sep 17;128(12):1335-40. doi: 10.1161/CIRCULATIONAHA.113.003059. Epub 2013 Aug 14. PMID 23946263
- [Derived] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to Cohort A if at least one stenoses had an FFR value of <=0.80. Participants with FFR >0.80 were treated according to local practice and were randomized to study follow-up / no study follow-up in Cohort B. Therefore, participants are either in cohort A or cohort B (not both).
Groups:
- Cohort A - PCI Plus OMT: PCI plus optimal medical treatment
  Stenting plus OMT: FFR guided PCI, plus OMT
- Cohort A - OMT Alone: Optimal medical treatment alone
  Standard of care: OMT alone
- Cohort B - Follow-up: Observation with treatment based on physician preference
- Cohort B - No Follow-up Re-consented: Observation with treatment based on physician preference, initially randomized to no follow-up, re-consented per safety data
Period: Overall Study
Arm/Group | Cohort A - PCI Plus OMT | Cohort A - OMT Alone | Cohort B - Follow-up | Cohort B - No Follow-up Re-consented
Started | 447 | 441 | 166 | 116
Completed | 407 | 403 | 146 | 104
Not Completed | 40 | 38 | 20 | 12
Not completed — Various reasons | 40 | 38 | 20 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - PCI Plus OMT | Cohort A - OMT Alone | Cohort B - Follow-up | Cohort B - No Follow-up Re-consented | Total
Number analyzed (Participants) | 447 | 441 | 166 | 116 | 1170
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.3) | 63.9 (9.6) | 63.6 (9.8) | 64.4 (8.8) | 63.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 103 | 53 | 37 | 286
  Male | 354 | 338 | 113 | 79 | 884

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac Event Rate (MACE)
Description: MACE: A composite of all cause death, documented MI, unplanned hospitalization leading to urgent revascularization.
Time Frame: 24 Month
Population: The primary outcome analysis was designed for Cohort A only.
Measure: Number; unit: percentage of subjects with SAEs
Groups:
- Cohort A - PCI Plus OMT: PCI plus optimal medical treatment - Stenting plus OMT: FFR guided PCI, plus OMT
- Cohort A - OMT Alone: Optimal medical treatment alone - Standard of care: OMT alone
Arm/Group | Cohort A - PCI Plus OMT | Cohort A - OMT Alone
Number analyzed (Participants) | 447 | 441
percentage of subjects with SAEs
  Non Urgent Revascularization | 6.7 | 32.7
  Death or Myocardial Infarction | 9.4 | 12.2
  Myocardial Infarction | 6.7 | 9.3
  Unplanned Hospitalizations with urgent revasc | 1.8 | 13.4
  Death | 3.6 | 3.9
  Cerebrovascular Event | 2.2 | 1.4
  Other Serious Adverse Event (SAE) | 0.2 | 0.7

2. Secondary Outcome: Overall MACE
Description: Individual components of the primary end point, cardiac death, and nonurgent revascularization
Time Frame: 3 years
Population: For registry cohort B, 50% of the patients with an FFR >0.80 across all lesions were followed up in a registry, and therefore, cohort B group for 'No Follow-up Re-consented' arm had no follow-up result and was not included in the endpoint analysis.
Measure: Number; unit: percentage of subjects
Groups:
- Cohort A: PCI Plus OMT: Patient with at least one hemodynamically significant stenosis (FFR, ≤0.80)
  PCI plus optimal medical treatment
  Stenting plus OMT: FFR guided PCI, plus OMT
- Cohort A: OMT Alone: Patient with at least one hemodynamically significant stenosis (FFR, ≤0.80)
  Optimal medical treatment alone
  OMT: OMT alone
- Cohort B: Registry Cohort: Patients in whom all stenoses had an FFR >0.80 were entered into a registry
Arm/Group | Cohort A: PCI Plus OMT | Cohort A: OMT Alone | Cohort B: Registry Cohort
Number analyzed (Participants) | 447 | 441 | 166
percentage of subjects
  Overall MACE | 10.1 | 22 | 12.7
  Death from any cause | 2.7 | 3.6 | 3.0
  Myocardial infarction | 6.3 | 7.7 | 6.6
  Urgent revascularization | 4.3 | 17.2 | 6.6
  Any revascularization | 10.3 | 44.2 | 14.5
  Nonurgent revascularization | 6.3 | 30.2 | 9.0
  Cardiac death | 1.1 | 1.1 | 1.8

ADVERSE EVENTS:
Time Frame: Unanticipated adverse device effects (UADE), major adverse cardiac event (MACE), serious adverse event (SAE) and stent thrombosis will be monitored through subject withdrawal following 3 year study follow-up.
Description: Only Serious Adverse Events were collected in this study.
Arm/Group | Cohort A - PCI Plus OMT | Cohort A - OMT Alone | Cohort B - Follow-up | Cohort B - No Follow-up Re-consented
Serious Adverse Events (participants affected / at risk) | 137/447 | 324/441 | 55/166 | 28/116
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - PCI Plus OMT (N=447) | Cohort A - OMT Alone (N=441) | Cohort B - Follow-up (N=166) | Cohort B - No Follow-up Re-consented (N=116)
Non Urgent Revacularization (Vascular disorders) | 30 (32) | 144 (162) | 14 (18) | 10 (11)
Death or MI (Cardiac disorders) | 42 (48) | 54 (65) | 16 (18) | 7 (7)
Myocardial Infarction (Cardiac disorders) | 30 (32) | 41 (48) | 11 (12) | 3 (3)
Unplanned Hospitalization with Urgent Revascularization (Vascular disorders) | 8 (8) | 59 (63) | 6 (6) | 3 (4)
Death (General disorders) | 16 (16) | 17 (17) | 6 (6) | 4 (4)
Cerebrovascular Event (General disorders) | 10 (10) | 6 (7) | 2 (2) | 1 (1)
Other SAE (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less